CLINICAL TRIAL: NCT06503211
Title: Phase I Clinical Study on the Safety, Tolerability, and Efficacy of UTAA09 Injection in the Treatment of Recurrent or Refractory B-cell Non Hodgkin's Lymphoma
Brief Title: On the Safety, Tolerability, and Efficacy of UTAA09 Injection in the Treatment of Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCART-19-002
Record Dates: First submitted 2024-07-07; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Recurrent or Refractory B-cell Non Hodgkin's Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, B-Cell

STUDY DESIGN:
Intervention Model Description: UTAA09 injection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- B cell injection targeting CD19 chimeric antigen receptor (Experimental): UTAA09 Injection The subjects, who sign the informed consent forms and been screeneinclusion/exclusion criteria, will be assigned into 3 x 108~1 x 1010 CD19-CAR - γδT cells.
  Interventions: Biological: UTAA09 injection

INTERVENTIONS:
Biological: UTAA09 injection — The subjects, who sign the informed consent forms and been screeneinclusion/exclusion criteria, will be assigned into 3 x 108~1 x 1010 CD19-CAR - γδT cells.

SUMMARY:
The main research objective is to evaluate the safety, tolerability, and pharmacokinetic characteristics of UTAA09 cell preparation in the treatment of relapsed/refractory B-cell non Hodgkin's lymphoma patients. The secondary research objective is to explore the clinical efficacy of UTAA09 injection after administration and to explore the content of CD19 positive B cells in peripheral blood after UTAA09 injection administration.

DETAILED DESCRIPTION:
Single dose, single arm trial, exploring the initial 28 day safety and efficacy of the investigational drug.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in clinical studies;
2. ECOG score 0-1 points;
3. Histologically confirmed large B-cell lymphoma, follicular lymphoma, mantle cell lymphoma, and inert lymphoma transformed into diffuse large B-cell lymphoma; CD19 and/or CD20 positivity;
4. At least one measurable tumor lesion determined according to Lugano's criteria: the longest diameter of intranodal lesions>1.5cm, and the longest diameter of extranodal lesions>1.0cm.

Exclusion Criteria:

1. Received other chimeric antigen receptor therapy or gene modified cell therapy before screening;
2. Subjects who were undergoing systemic steroid therapy during screening and were determined by the researchers to require long-term use of systemic steroid therapy during the treatment period (excluding inhalation or local use);
3. Any unstable heart disease, including but not limited to unstable angina, myocardial infarction (within 6 months prior to screening), congestive heart failure (New York Heart Association [NYHA] classification ≥ III), and severe arrhythmia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-07-31 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of dose limiting toxicity (DLT ) | 28 days after infusion
  The incidence, severity, and types of dose limiting toxicity
The incidence of TEAEs | 28 days after infusion
  The incidence, severity, and types of adverse events that occur during treatment

SECONDARY OUTCOMES:
ORR | 24 months after infusion
  Evaluate the overall response rate based on the efficacy criteria of Lugano 2014
PFS | 24 months after infusion
  Evaluate the progression free survival based on the efficacy criteria of Lugano 2014
OS | 24 months after infusion
  Evaluate the overall survival based on the efficacy criteria of Lugano 2014

CONTACTS AND LOCATIONS:
Overall Officials: Xu Huang, Bachelor, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- PersonGen.Anke Cellular Therapeutice Co., Ltd., Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No